CLINICAL TRIAL: NCT06409520
Title: Impact Of Subclinical Hypothyroidism On Short-Term Outcomes In Patients With Acute Coronary Syndrome In Sohag University Hospitals
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amr Ibrahim Abd El-haleem Adam, Assistant lecturer internal medicine sohag university, Sohag University
Other Study IDs: soh-Med-24-04-04MD
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Subclinical hypothyroïdism; Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Thyroid Function Tests; Electrocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group (1): patients with acute coronary syndrome and subclinical hypothyroidism
  Interventions: Diagnostic Test: thyroid function tests; Diagnostic Test: cardiac enzymes; Diagnostic Test: ECG
- Group (2): (control group) patients with acute coronary syndrome and normal thyroid function
  Interventions: Diagnostic Test: thyroid function tests; Diagnostic Test: cardiac enzymes; Diagnostic Test: ECG

INTERVENTIONS:
Diagnostic Test: thyroid function tests — (TSH, free T4) The normal ranges of thyroid function tests were 0.40-4.99 mIU/L for TSH and 0.7-1.8 ng/dL for free T4. The same testing method will performed on all samples from all patients.
Diagnostic Test: cardiac enzymes — troponine
Diagnostic Test: ECG — Electrocardiogram

SUMMARY:
Introduction:

Subclinical hypothyroidism (SCH) is defined biochemically as a normal serum free thyroxine (T4) level in the presence of an increased serum thyroid stimulating hormone (TSH) concentration.(1) Its prevalence ranges from 4 to 15 percent and is higher in females and increasing age.(2) Overt hypothyroidism was associated with accelerated atherosclerosis and an increased risk of cardiovascular abnormalities. (3) Some studies have reported a higher atherosclerotic cardiovascular disease risk in patients with SCH. (5-8) Elevated TSH levels were observed to be associated with higher cholesterol levels.(9) Higher mortality was also reported in some studies (6,10) especially with TSH ≥ 10.0 mIU/L, in contrast to other studies.(11,12) Heart failure events and myocardial infarction have been reported to be higher.(13,14) These findings in SCH patients could be explained by mitochondrial oxidative stress due to elevated inflammatory markers, hypercoagulability, endothelial dysfunction, insulin resistance, increased vascular resistance and left ventricular diastolic and systolic dysfunction.(3,15,16) As is the case with overt hypothyroidism, SCH was observed to be associated with elevated peripheral vascular resistance and diastolic dysfunction.(17) There are a few studies evaluating the effects of subclinical hypothyroidism on the outcomes of acute coronary syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years) diagnosed with acute coronary syndrome

Exclusion Criteria:

1. Patients with overt hypothyroidism or hyperthyroidism.
2. Pregnant and lactating females
3. Patients with severe comorbid conditions e.g. Malignancy decompensated liver diseases or end stage kidney diseases.
4. Patients with a history of taking medications affecting thyroid function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (age ≥18 years) diagnosed with acute coronary syndrome
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Short-term complications | 1 year
  events during hospitalisation will be documented, and patients will be followed up for 30 days. The documented inhospital events include cardiogenic shock, Ejection fraction less than 40%, Killip class more than one, new atrial fibrillation, sudden cardiac arrest, bradyarrhythmia necessitating pacing, major bleeding necessitating blood transfusion, and acute kidney injury while hospitalized

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cooper DS, Biondi B. Subclinical thyroid disease. Lancet. 2012 Mar 24;379(9821):1142-54. doi: 10.1016/S0140-6736(11)60276-6. Epub 2012 Jan 23. PMID 22273398
- [Background] Sun J, Yao L, Fang Y, Yang R, Chen Y, Yang K, Tian L. Relationship between Subclinical Thyroid Dysfunction and the Risk of Cardiovascular Outcomes: A Systematic Review and Meta-Analysis of Prospective Cohort Studies. Int J Endocrinol. 2017;2017:8130796. doi: 10.1155/2017/8130796. Epub 2017 Aug 31. PMID 29081800
- [Background] Inoue K, Ritz B, Brent GA, Ebrahimi R, Rhee CM, Leung AM. Association of Subclinical Hypothyroidism and Cardiovascular Disease With Mortality. JAMA Netw Open. 2020 Feb 5;3(2):e1920745. doi: 10.1001/jamanetworkopen.2019.20745. PMID 32031647
- [Background] Hyland KA, Arnold AM, Lee JS, Cappola AR. Persistent subclinical hypothyroidism and cardiovascular risk in the elderly: the cardiovascular health study. J Clin Endocrinol Metab. 2013 Feb;98(2):533-40. doi: 10.1210/jc.2012-2180. Epub 2012 Nov 16. PMID 23162099
- [Background] Suh S, Kim DK. Subclinical Hypothyroidism and Cardiovascular Disease. Endocrinol Metab (Seoul). 2015 Sep;30(3):246-51. doi: 10.3803/EnM.2015.30.3.246. Epub 2015 Aug 4. PMID 26248862